CLINICAL TRIAL: NCT04956172
Title: Assessing the Impact of the NeuroCatch Platform 2 Stimulus Tone Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NCI_NCClin_005
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Brain Health

STUDY DESIGN:
Intervention Model Description: This is a within-subject repeated-measures, randomly counterbalanced, single blind study.
  All participants will be asked to attend two study visits, one week (6-8 days) apart. At each study visit, participants will complete two NeuroCatch Platform 2 assessments with different auditory sequences. One sequence will include the Standard Tone A (80dB), and another will include Standard Tone B (93dB) while keeping the deviant tone volume consistent (105dB). The order of presentation of the two sequences will be randomly counterbalanced (i.e Session 1: AB & Session 2: BA, or Session 1: BA & Session 2: AB).
Who Masked: Participant
Masking Description: Participants are not informed the order or type (standard Tone A, standard Tone B) of the sequences
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tone A (Active Comparator): Tone A uses an 80dB standard tone
  Interventions: Device: NeuroCatch Platform 2
- Tone B (Experimental): Tone B uses a 93dB standard tone
  Interventions: Device: NeuroCatch Platform 2

INTERVENTIONS:
Device: NeuroCatch Platform 2 — To elicit the ERP components of interest in this study (N100, P300, N400), proprietary auditory stimulus sequences will be administered using the NeuroCatch Platform 2, an investigational medical device. Each sequence consists of tones and word pairs to elicit the various components of interest. The NeuroCatch Platform 2 consists of a computerized acquisition software which presents the stimulus, acquires the data and presents the amplitude and latency values of the ERP components (N100, N400, P300)

SUMMARY:
The NeuroCatch Platform 2 (NCP2), an investigational medical device system developed by NeuroCatch Inc., consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP; brain response to a stimulus) information.

The NCP2 uses two types of tones to elicit N100 and P300 ERPs, along with two types of words to elicit N400 ERPs. The objective of this study is to determine if changing the volume of the standard tone has an effect on the amplitudes and latencies of the ERPs.

DETAILED DESCRIPTION:
Electroencephalography (EEG) signals have been collected and studied since the early 1970s as a non-invasive way of assessing brain function. As early as the 1930s, a derivative of the raw EEG signal - event-related potentials (ERPs) - were computed. These scalp-recorded ERPs are the brain's response to a stimulus of interest (e.g. a flashing checkerboard or an angry face). The size, timing, and topographical location of ERP components lend insight into the timing and complexity of various cognitive processes. At NeuroCatch Inc. (NCI), research is primarily focused on three ERP components: the N100, P300 and N400, associated with different attention abilities (sensory processing, target detection & semantic processing).

The N100 is a negative-going deflection around 100 ms post stimulus onset. This particular ERP component indexes sensory stimulus at a pre-attentive level, or in other words, the acknowledgement by the brain that information has entered the system. Whereas the P300 - a positive-going deflection around 300 ms - indexes an early stage of attentional processing. This component is particularly sensitive to context updating or target identification (the brain's 'Ah-ha!' response). Finally, the N400 is a negative-going deflection peaking around 400 ms post stimulus. This component is measured in situations of semantic violations (e.g. 'The pizza was too hot to … lamp"), thus indexing one of the highest-order cognitive functions: language processing.

Each of the three ERP components have been studied in academic laboratories for multiple decades and prototypical values for their timing (latency) and size (amplitude) have become widely accepted. To elicit the ERP components of interest in this study (N100, P300, N400), proprietary auditory stimulus sequences will be administered using the NeuroCatch Platform 2, an investigational medical device. Each sequence consists of tones and word pairs to elicit the various components of interest. Standard tones (lower volume, low pitch) make up most of the tones in the sequence, with deviant tones (higher volume, higher pitch) inserted in random intervals. The difference in volume and pitch between the standard tones and deviant tones, coupled with the "unexpected" nature of the deviant tone, is what drives the N100 and P300 responses.

NeuroCatch Platform 2 consists of a computerized acquisition software which presents the stimulus, acquires the data and presents the amplitude and latency values of the ERP components (N100, N400, P300). This protocol is intended to assess the effect of changing the standard tone volume in the NeuroCatch Platform 2 auditory tone sequences on the elicited ERP responses.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex, at least 19 years of age or older
2. Able to understand the informed consent form, study procedures and willing to participate in study
3. Able to remain seated and focused for 7 minutes
4. In good health with no history of clinically relevant neurological illness or injury in the last 5 years

Exclusion Criteria:

1. Requires the use of hearing aids or a cochlear implant, diagnosed with tinnitus that is currently active, or has temporary damage to hearing (e.g. punctured ear drum).
2. Implanted pacemaker or implanted electrical stimulators
3. Metal or plastic implants in the skull, excluding dental/facial implants.
4. Exposed to an investigational drug or device 30 days prior to start in this study, or concurrent or planned use of investigational drug or device while enrolled in this study
5. Not proficient in English language
6. Diagnosed epilepsy or history of seizures
7. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
8. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin)
9. Allergy to EEG gel or history of contact dermatitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in amplitude of the N100 ERP | 1 week (6-8 days)
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the difference in amplitude between the two Tone types will be a full-factorial repeated measures analysis of variance (Factors: Tone type, Session number, Run number)
Difference in latency of the N100 ERP | 1 week (6-8 days)
  Latency (response time) will be measured in microseconds. The statistic being used to measure the difference in amplitude between the two Tone types will be a full-factorial repeated measures analysis of variance (Factors: Tone type, Session number, Run number)
Difference in amplitude of the P300 ERP | 1 week (6-8 days)
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the difference in amplitude between the two Tone types will be a full-factorial repeated measures analysis of variance (Factors: Tone type, Session number, Run number)
Difference in latency of the P300 ERP | 1 week (6-8 days)
  Latency (response time) will be measured in microseconds. The statistic being used to measure the difference in amplitude between the two Tone types will be a full-factorial repeated measures analysis of variance (Factors: Tone type, Session number, Run number)
Difference in amplitude of the N400 ERP | 1 week (6-8 days)
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the difference in amplitude between the two Tone types will be a full-factorial repeated measures analysis of variance (Factors: Tone type, Session number, Run number)
Difference in latency of the N400 ERP | 1 week (6-8 days)
  Latency (response time) will be measured in microseconds. The statistic being used to measure the difference in amplitude between the two Tone types will be a full-factorial repeated measures analysis of variance (Factors: Tone type, Session number, Run number)

SECONDARY OUTCOMES:
Repeatability of the N100 Amplitude for Tone A | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the N100 Amplitude for Tone B | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the N100 Latency for Tone A | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the N100 Latency for Tone B | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the P300 Amplitude for Tone A | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the P300 Amplitude for Tone B | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the P300 Latency for Tone A | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the P300 Latency for Tone B | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the N400 Amplitude for Tone A | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the N400 Amplitude for Tone B | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the N400 Latency for Tone A | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Repeatability of the N400 Latency for Tone B | 1 week (6-8 days)
  The statistic being used to measure the repeatability will be the two-way mixed single measures absolute agreement type of intraclass correlation coefficient (denoted as ICC(A,1)
Collection and evaluation of adverse events and adverse device effects | At time of event
  Evaluation of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Bimal Lakhani, PhD, Study Chair — NeuroCatch Inc.
Locations (1):
- HealthTech Connex Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided